CLINICAL TRIAL: NCT01273740
Title: Swedish External Support Study is Randomized Trial of the Effect of External Support of PTFE-grafts for Bypass to Below Knee Arteries.
Brief Title: Swedish External Support Study
Acronym: SWEXSUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Lasarettet Boden (Other); Borås Lasarett (Other); Eskilstuna Lasarettet (Other); Falu Lasarett Röntgen (Other); Department of Surgery, Sahlgrenska sjukhuset, Göteborg (Unknown); Department of Surgery, Östra sjukhuset, Göteborg (Unknown); Lasarett Gävle (Other); Helsingborgs Hospital (Other); Kalmar County Hospital (Other); Karlstad Central Hospital (Other); Kristiansund Hospital (Other); Lund University Hospital (Other); Malmö University (Other); Department of Surgery, Lasarettet, Motala (Unknown); Department of Surgery, Lasarettet, Mölndal (Unknown); Department of Surgery, Lasarettet, Norrköping (Unknown); Department of Surgery, Lasarettet, Nyköping (Unknown); Department of Surgery, Lasarettet, Skellefteå (Unknown); Department of Surgery, Kärnsjukhuset, Skövde (Unknown); Department of Surgery, S:t Görans Sjukhus, Stockholm (Unknown); Department of Surgery, Södersjukhuset, Stockholm (Unknown); Department of Surgery, Norra Älvsborgs Länssjukhus, Trollhättan-Vänersborg (Unknown); Uppsala University Hospital (Other); Västervik Hospital (Other); Region Västmanland (Other); Department of Surgery, Lasarettet, Växjö (Unknown); Department of Surgery, Lasarettet, Örebro (Unknown); Department of Surgery, Lasarettet, Östersund (Unknown)
Responsible Party: Fredrik Lundgren, Department of CardioVascylar Surgery, Universityhospital, Linköping, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWEXSUS
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Critical Limb Ischemia
Keywords: PTFE bypass; femoro-popliteal; femoro-crural; popliteal arteries; crural arteries; external support; crtical limb ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- External support (Experimental): Bypass graft with external support
  Interventions: Procedure: External support
- No external support (Experimental): Bypass with graft without external support
  Interventions: Procedure: External support

INTERVENTIONS:
Procedure: External support — Bypass surgery with externally supported graft

SUMMARY:
Randomized study to evaluate the effect of adding external support to PTFE-grafts used for bypass to below knee arteries in patients with critical limb ischemia with respect to primary patency, secondary patency, and limb salvage.

ELIGIBILITY:
Inclusion Criteria:

Critical limb ischemia Need for bypass surgery

Exclusion Criteria:

Can participate in follow-up Has suitable saphenous vein

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 1995-01; Primary Completion 1998-06 (Actual); Study Completion 1998-06 (Actual)

PRIMARY OUTCOMES:
primary graft patency

SECONDARY OUTCOMES:
limb salvage

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik BG Lundgren, PhD, MD, Principal Investigator — Department of CardioVascular Surgery, University Hospital, Linköping, Sweden